CLINICAL TRIAL: NCT03845608
Title: Postoperative Analgesic Efficacy of the Pulmonary Recruitment Maneuver Compared to Intraperitoneal Hydrocortisone in Laparoscopic Gynecological Surgery
Brief Title: Analgesic Effect of Pulmonary Recruitment and Intraperitoneal Hydrocortisone in Laparoscopic Gynecological Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: pain and laparoscopic surgery
Record Dates: First submitted 2018-09-29; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Laparoscopic Gynecological Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary Recruitment Maneuver (Experimental): Pulmonary recruitment maneuver will be performed manually using positive-pressure ventilation to inflate the lungs and lower the diaphragm, which can increase intraperitoneal pressure mechanically and remove residual carbon dioxide from the peritoneal cavity
  Interventions: Combination Product: Pulmonary Recruitment Maneuver
- Intraperitoneal Hydrocortisone (Other): Drug Injection: 100mg of Hydrocortisone will be injected In the peritoneum
  Interventions: Combination Product: Pulmonary Recruitment Maneuver
- control group (No Intervention): In the controls, carbon dioxide will be removed by the traditional passive deflation of abdominal cavity.

INTERVENTIONS:
Combination Product: Pulmonary Recruitment Maneuver — Pulmonary recruitment maneuver will be performed manually using positive-pressure ventilation to inflate the lungs and lower the diaphragm, which can increase intraperitoneal pressure mechanically and remove residual carbon dioxide from the peritoneal cavity.recieve100 mg hydrocortisone in 250 ml normal saline at end of surgery and carbon dioxide will be removed by applying gentle abdominal pressure and removing carbon dioxide by passive exsufflation
  Arms: Intraperitoneal Hydrocortisone; Pulmonary Recruitment Maneuver

SUMMARY:
The aim of this study is to compare the postoperative analgesic efficacy of intraperitoneal hydrocortisone to pulmonary recruitment maneuver in Laparoscopic gynaecological surgery.

DETAILED DESCRIPTION:
Laparoscopic surgeries are becoming more attractive because of an early recovery . However, post laparoscopic shoulder and upper abdominal pain may cause more discomfort to the patient than the pain at the incision site.

Proper pain relief is a major concern and area of focus. Pre-operatively, one of the most common questions asked by patients about the amount of pain they will experience after the surgery. Pain has been found to be one of the three most common medical causes of delayed discharge after ambulatory surgery, the other two being drowsiness and nausea and vomiting. Unfortunately prevention and treatment of postoperative pain continues to be a major challenge in postoperative care.

Good pain control after surgery is important to prevent negative outcomes such as tachycardia, hypertension, myocardial ischemia, decrease in alveolar ventilation, and poor wound healing.

Pain also can prolong hospital stay, which is particularly important in day case procedures.

The mechanism of laparoscopy induced shoulder pain is mainly derived from carbon dioxide retention within the abdomen, subsequently irritating the phrenic nerve and causing referred pain in the C4 dermatome. Moreover, carbon dioxide trapped between the liver and the right diaphragm, irritating the diaphragm, also causes upper abdominal pain.

Although there are many analgesic drugs available for postoperative pain, many patients still find them to be suboptimal for controlling pain.

Many strategies, including treatment with non steroidal anti-inflammatory drugs, have been used to try to reduce laparoscopy-induced shoulder pain however, no sufficiently reliable methods have been reported yet .

Also Intraperitoneal local anesthetic was tried as an important addition for postoperative pain in the era of modern surgery. The method of delivering local anesthetic directly to the intraperitoneal cavity was first described in 1951 by Griffin et al. ; however, this method was forgotten for many years until its implementation in minimal access surgery was reappeared. It significantly reduces postoperative pain and opioid consumption after laparoscopic gynecological and general surgical operations.

Another effective method is the pulmonary recruitment maneuver (PRM) which can mechanically remove residual carbon dioxide and therefore decreasing peritoneal irritation, and shoulder pain.

Intravenous steroids have been used successfully for postoperative pain relief in different kinds of surgery . Also intraperitoneal hydrocortisone was has been used effectively to reduce pain after laparoscopic cholecystectomy.

In addition combination of intraperitoneal local anesthetics with hydrocortisone was proved to be a successful method in controlling upper abdominal and shoulder pain after laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* • female gender, age 20-45 years undergoing laparoscopic gynecological operations

  * American Society of Anesthesiologist physical status classification of I or II

Exclusion Criteria:

* • Patients younger than 20 years or older than 45 years

  * History of chronic pain
  * Regular medication with analgesics, or steroids
  * Analgesic use within 24 h of surgery ,drug or alcohol abuse
  * Associated chronic diseases like diabetes mellitus, pulmonary diseases ,poor cardiac reserve,hepatorenal insufficiency.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The first 24 hours total analgesic consumption. | 24 hours after surgery
  Total amount of opioid drugs used after surgery for assessment of post operative pain

SECONDARY OUTCOMES:
Length of the recovery and hospital stay (hours) | 24 hours postoperative
  Duration between end of operation and patient discharge from hospital
Incidence of postoperative nausea ,vomiting or abdominal distension(%) | 24 hours postoperative
  gastrointestinal complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nesrine El-Refai, MD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kluivers KB, Johnson NP, Chien P, Vierhout ME, Bongers M, Mol BW. Comparison of laparoscopic and abdominal hysterectomy in terms of quality of life: a systematic review. Eur J Obstet Gynecol Reprod Biol. 2008 Jan;136(1):3-8. doi: 10.1016/j.ejogrb.2007.06.004. Epub 2007 Dec 11. PMID 18063290
- [Background] Vadivelu N, Mitra S, Narayan D. Recent advances in postoperative pain management. Yale J Biol Med. 2010 Mar;83(1):11-25. PMID 20351978
- [Background] Jackson SA, Laurence AS, Hill JC. Does post-laparoscopy pain relate to residual carbon dioxide? Anaesthesia. 1996 May;51(5):485-7. doi: 10.1111/j.1365-2044.1996.tb07798.x. PMID 8694166
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Background] Kahokehr A. Intraperitoneal local anesthetic for postoperative pain. Saudi J Anaesth. 2013 Jan;7(1):5. doi: 10.4103/1658-354X.109554. No abstract available. PMID 23717222
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Background] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749
- [Background] Safavi M, Honarmand A, Habibabady MR, Baraty S, Aghadavoudi O. Assessing intravenous ketamine and intravenous dexamethasone separately and in combination for early oral intake, vomiting and postoperative pain relief in children following tonsillectomy. Med Arh. 2012;66(2):111-5. doi: 10.5455/medarh.2012.66.111-115. PMID 22486143